CLINICAL TRIAL: NCT00709033
Title: Phase I Study Of The Administration Of Peripheral Activated T-Cells and EBV Specific CTLs Expressing CD19 Chimeric Receptors For Advanced B-Cell Non-Hodgkin's Lymphoma And Chronic Lymphocytic Leukemia (ATECRAB)
Brief Title: T-cells or EBV Specific CTLs, Advanced B-Cell NHL and CLL
Acronym: ATECRAB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22899-ATECRAB; ATECRAB (Other: Baylor College of Medicine)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: refractory; relapsed; low; intermediate-grade; Non-Hodgkin lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- autologous or syngeneic PBTLs and EBV-CTLs (Experimental): The subject will be assigned a dose of CD19-CD28 chimeric receptor T cells at study entry.
  Interventions: Biological: autologous or syngeneic PBTLs and EBV-CTLs

INTERVENTIONS:
Biological: autologous or syngeneic PBTLs and EBV-CTLs — Three dose levels are being evaluated namely:
  GROUP 1
  PBTL CD19CAR-28 zeta 2x10exp7 cells/m2 and EBV-CTL CD19CAR zeta 2x10exp7 cells/m2
  GROUP 2
  PBTL CD19CAR-28 zeta 1x10exp8cells/m2 and EBV-CTL CD19CAR zeta 1x10exp8 cells/m2
  GROUP 3
  PBTL CD19CAR-28 zeta 2x10exp8 cells/m2 and EBV-CTL CD19CAR zeta 2x10exp8 cells/m2

SUMMARY:
Patients on this study have a type of lymph gland cancer called non-Hodgkin Lymphoma or chronic Lymphocytic Leukemia. Their lymphoma or CLL has come back or has not gone away after treatment. Because there is no standard treatment for the cancer at this time or because the currently used treatments do not work fully in all cases, patients are being asked to volunteer to take part in a gene transfer research study using special immune cells.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise, but have not been strong enough to cure most patients.

The antibody used in this study is called anti-CD19. This antibody sticks to lymphoma cells because of a substance on the outside of these cells called CD19. CD19 antibodies have been used to treat people with lymphoma and CLL. For this study, the anti-CD19 antibody has been changed so that instead of floating free in the blood it is now attached to T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These chimeric receptor-T cells seem to be able to kill tumors, but they don't last very long and so their chances of fighting the cancer are limited.

Investigators found that T cells work better if they also attach a protein called CD28 to the T cells. This protein makes the T cells more active and survive longer.

Also they found that T cells that are also trained to recognize the virus that causes infectious mononucleosis (called Epstein Barr Virus or EBV) can stay in the blood stream for many years.

These CD19-CD28 chimeric receptor T cells and CD19 chimeric-EBV specific T cells are investigational products not approved by the FDA.

The purpose of this study is to find the biggest dose of chimeric T cells that is safe to administer, to see how long each of the T cell populations (CD19-CD28 and CD19-EBV-specific) last, to assess what the side effects are, and to evaluate whether this therapy might help people with lymphoma or CLL.

DETAILED DESCRIPTION:
The patient or their donor will give us blood to make CD19-CD28 chimeric receptor T cells and CD19 chimeric-EBV specific T cells in the laboratory. These cells are grown and frozen for the patient. Because the patient will have received cells with a new gene in them they will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

The patient will be assigned a dose of CD19-CD28 chimeric receptor-T cells and CD19 chimeric receptor-EBV specific T cells. Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in circulation. Because of that, if the patient's level of circulating T cells is relatively high, they will receive one treatment of cyclophosphamide. This drug will decrease the numbers of the patient's own T cells before the infusion the CD19 chimeric receptor T cells. Although it's not expected to have any effect on the tumor with the dose that the subject will receive, this drug is part of many regimens that are used to treat lymphoma or CLL. If the subject is already receiving chemotherapy, this may not be needed.

The patient will be given an injection of cells into the vein through an IV line at the assigned dose. The patient will be followed in the clinic after the injection for up to 3 hours. If after a 4-6 week evaluation period after the infusion, the patient seems to be experiencing a benefit (confirmed by radiological studies, physical exam and/or symptoms), they may be able to receive up to three additional doses of the T cells. These additional infusions would be at least 4-6 weeks apart and at the same dose level the patient received the first time.

ELIGIBILITY:
INCLUSION CRITERIA:

FOR TREATMENT:

* Recurrent low or intermediate grade B-cell lymphoma or B-CLL, or newly diagnosed patients unable to receive or complete standard therapy OR diagnosis of relapsed/refractory intermediate B cell lymphoma with a treatment plan that will include high dose therapy and autologous stem cell transplantation.
* CD19-positive tumor
* EBV seropositivity (in patient and donor, as applicable)
* Recovered from the acute toxic effects of all prior chemotherapy at least a week before entering this study.
* Not be currently receiving any investigational agents or have not received any tumor vaccines within the previous six weeks.
* No treatment with rituximab within the previous 8 weeks.
* ANC > 500, Hgb > 8.0*
* Bilirubin less than 3 times the upper limit of normal*
* AST less than 5 times the upper limit of normal*
* Serum creatinine less than 3 times upper limit of normal*
* Pulse oximetry of > 90% on room air*
* Adequate pulmonary function with FEV1, FVC and DLCO >35%* of expected corrected for hemoglobin
* Karnofsky or Lansky score of > 60%.
* Available autologous or syngeneic transduced EBV-specific cytotoxic T lymphocytes and peripheral blood T-cells with 15% or greater expression of CD19CAR determined by flow-cytometry.
* Patients or legal guardians must understand and sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 3 months after the study is concluded. The male partner should use a condom.

EXCLUSION CRITERIA:

* History of hypersensitivity reactions to murine protein-containing products.
* Pregnant or lactating.
* Tumor in a location where enlargement could cause airway obstruction.
* Active infection with HIV, HBV, HCV or CMV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity | 6 weeks
  Dose-limiting toxicity is defined as development of NCI grade III - IV non-hematologic or grade IV hematologic toxicity that can be attributed to the study treatment

SECONDARY OUTCOMES:
Survival and function of CD19CAR PBTLs and EBV-CTLs | 15 years
  To measure the differential survival and function of CD19CAR transduced PBTLs and EBV-CTLs in vivo, in particular to determine if CD19CAR transduced EBV-CTLs survive longer than CD19CAR-CD28 transduced PBTLs.
Number of patients with tumor response | 6 weeks
  To measure the anti-tumor effects of CD19CAR transduced T- lymphocytes in patients with low and intermediate-grade NHL or B-CLL.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Xu Y, Zhang M, Ramos CA, Durett A, Liu E, Dakhova O, Liu H, Creighton CJ, Gee AP, Heslop HE, Rooney CM, Savoldo B, Dotti G. Closely related T-memory stem cells correlate with in vivo expansion of CAR.CD19-T cells and are preserved by IL-7 and IL-15. Blood. 2014 Jun 12;123(24):3750-9. doi: 10.1182/blood-2014-01-552174. Epub 2014 Apr 29. PMID 24782509

DOCUMENTS (1):
  • Informed Consent Form (2013-05-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT00709033/ICF_000.pdf